CLINICAL TRIAL: NCT02656108
Title: Omission of Controlled Cord Traction During Active Management of Third Stage of Labor. A Single Blinded Randomized Controlled Trial
Brief Title: Omission of Controlled Cord Traction During Active Management of Third Stage of Labor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed El Kotb Abdel Fattah, dr. Ahmed Kotb, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CCO
Record Dates: First submitted 2016-01-12; First posted 2016-01-14 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Labor Stage, Third

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- omiited controlled cord traction (Experimental): neither controlled cord traction nor fundal pressure will be applied. The placenta will be delivered physiologically and signs of placental separation will be awaited
  Interventions: Procedure: Ommited controlled cord traction
- controlled cord traction (Active Comparator): the cord will be held in one hand and the other hand will be placed just above the woman's pubic boneto stabilize the uterus during cord traction
  Interventions: Procedure: controlled cord traction

INTERVENTIONS:
Procedure: Ommited controlled cord traction — No controlled cord traction and no fundal pressure. placenta will be allowed to deliver physiologically
  Arms: omiited controlled cord traction
Procedure: controlled cord traction — active management of third stage of labor in the form of uterine massage with controlled cord traction
  Arms: controlled cord traction

SUMMARY:
This is a comparative study which will be conducted in Ain Shams University Maternity hospital to assess the individual and specfic role of controlled cord traction as a part of active management of third stage of labor

DETAILED DESCRIPTION:
300 patients will be randomized into two groups with controlled cord traction and withoout. The primary outcome will be sever postpartum haemorrhage

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* term pregnancy

Exclusion Criteria:

* episiotomy
* operative vaginal delivery
* known coagulation defect
* Acute complication during labor e.g. eclampsia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 320 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
sever post partum haemorrhage | 24 hours
  blood loss more than 500 cc

SECONDARY OUTCOMES:
duration of third stage of labor | 30 minutes
  from delivery of the baby to delivery of the placenta

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M kotb, MD, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No